CLINICAL TRIAL: NCT06718803
Title: A Mobile App for Hot Flashes and Sleep Disturbances (Evia): Randomized Controlled Trial
Brief Title: A Mobile App for Hot Flashes and Sleep Disturbances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Responsible Party: Principal Investigator, Vanessa Muniz, Principal Investigator, Baylor University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2220078
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Hot Flashes
Keywords: Hypnosis; post-menopausal; mhealth; apps; hypnotherapy; hot flashes
MeSH Terms: conditions — Hot Flashes | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hypnotherapy App (Experimental): Participants in the experimental arm will be asked to engage with a mobile health app that provides hypnotherapy and educational resources tailored for managing hot flashes. The hypnotherapy app offers a structured 5-week program adapted from a hypnosis protocol that has been tested in various randomized clinical trials (Elkins et al., 2008; Elkins et al., 2013). During the 5-week program, users engage in daily activities such as reading brief educational materials, undergoing hypnotic sessions, and tracking their hot flashes. The app also offers users with optional hypnotherapy to improve sleep quality. The hypnotherapy app uses audio recordings to deliver hypnotherapy remotely, these are composed of mental imagery techniques focused on sensations of coolness, such as imagining cool breezes, snow, and a sense of calmness.
  Interventions: Behavioral: Hypnosis
- Health and habits tracker app (Placebo Comparator): Participants assigned to the comparator group will be asked to engage with a daily health and habits tracker app, participants will access the control app free-of-charge, and will be asked to use the app for the five-week period. The app provides users with an interface that facilitates tracking of symptoms, physical activity, medications, and more. Participants will be asked to track their number of hot flashes, sleep quality, and additional symptoms and habits related to the management of hot flashes. Instructions regarding suggestions on what to track and how to maximize app usage will be provided to the participants by our research coordinator. Data will not be collected from the app.

INTERVENTIONS:
Behavioral: Hypnosis — The Evia program includes three mayor components, 1. A hypnotherapy program for the reduction of hot flashes, 2. Educational readings on hot flashes and menopausal-related topics, 3. Daily hot flash tracker.
  The hypnotherapy is delivered in short, daily 10-20 minute audio recordings that involve numerous suggestions for coolness and relaxation (i.e., cool breeze, snowy mountain, deep lake) for a period of five weeks. The hypnotherapy program is based on previous randomized controlled trials for the reduction of hot flashes (Elkins et al., 2008; Elkins et al., 2013).
  Other Names: hypnotherapy; hypnotic relaxation therapy; clinical hypnosis
  Arms: Hypnotherapy App
Other: Structured Attention — Data collection of hot flash severity and frequency will mirror the hot flashes daily tracker offered by the intervention group (Evia app), and account for time and structured attention control while removing any potential therapeutic effects.

SUMMARY:
The purpose of the study is to compare the possible efficacy and acceptability of two mobile health applications for the reduction of hot flashes and related symptoms.This study is completely remote, and participants will be be asked to engage with a mobile health application daily for five weeks and provide feedback and experience with the app.

DETAILED DESCRIPTION:
The North American Menopause Society's 2023 position statement on non-hormonal interventions for hot flashes has recognized hypnotherapy as a Level 1 recommended intervention, meaning there is good and consistent scientific evidence for the intervention. Hypnotherapy for hot flashes has been shown to be an efficacious treatment for hot flashes (hot flashes measured by hot flash daily diaries and the Hot Flash Related Daily Interference Scale) when administered face-to-face, with women experiencing on average between 70% reductions in hot flashes, which is well over the clinically significant threshold of 50% reduction. In addition, hypnotherapy for hot flashes has been shown to improve sleep quality by up to 50% on average.

Further, a mobile app (Evia) has been developed by Mindset Health to deliver hypnotherapy for hot flashes. Evia is an app that delivers a 5-week program for hypnotic inductions and educational information for hot flashes. The app provides daily tasks such as educational readings, hypnotic inductions, and tracking hot flashes. Due to growth in smartphone ownership and an increase in remotely delivered mobile health (mHealth) apps for smartphones, it is clear that smartphone apps are a strategic way to increase access to hypnosis interventions for hot flashes.

However, there has not yet been a randomized controlled trial evaluating the mobile app for hot flash reduction in menopausal women. The goal of this feasibility randomized clinical trial study is to evaluate the feasibility and potential efficacy of hypnotherapy delivered through the use of a mHealth app vs. a daily health and habit-tracker app for the reduction of hot flashes and improved sleep quality. This proposal delineates three specific aims.

Aim 1: To assess the feasibility of remote accrual of menopausal women with at least 36 weekly hot flashes, randomization to both apps, and retention.

Aim 2: To assess the feasibility of data collection, and the potential efficacy of hypnotherapy on primary and secondary outcomes (i.e., hot flash diaries, interference caused by hot flashes, physiologically-measured hot flash frequency, sleep quality, anxiety, heart palpitations, stress).

Aim 3: To evaluate the satisfaction rating and adverse events. After using the apps for 5 weeks, participants will provide satisfaction ratings on a 0-10 scale (0=completely unsatisfied and 10=completely satisfied. We will also inquire about and record any reported adverse events related to or unrelated to the use of this study's apps.

Aim 4: To explore the feasibility of measuring hypnotizability and practice adherence in a completely remote, mhealth app-based study.

ELIGIBILITY:
Inclusion Criteria:

* 40 years or older and able to consent to participate in the study.
* Self-reported history of a minimum of 36 hot flashes per week at baseline.
* Ability to access the app to which the participant is randomized to (the Evia app or the Talli Care app).
* Ability to speak and understand English. Non-English speakers are not considered in this study because the Apps are currently only offered in English.

Exclusion Criteria:

* New or changes in the current use of any prescription or complementary and alternative medicine (CAM) treatments for hot flashes during the duration of the intervention. [If the participant is already using any prescription or CAM, they will be asked to provide details of ingredients, dose and frequency. They will be permitted to participate in the study if they agree to no change for the duration of their participation in the study and otherwise meet inclusion criteria.]
* Does not have access to a Smartphone
* Severe or unstable medical or psychiatric illness.
* Current use of hypnosis for any condition.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Hot Flash Daily Diaries | From enrollment to the end of treatment (week 6)
  Hot flash frequency and hot flash scores will be measured using hot flash daily diaries (Sloan et al., 2001) to assess the feasibility of the intervention for the reduction of hot flashes compared to a structured attention control condition. Hot flash daily diaries are a reliable measure of hot flash frequency and severity most commonly used in prior randomized control trials using hypnotherapy for hot flash treatment (Barton et al., 2017; Elkins et al., 2008; Elkins et al., 2013; MacLaughlan et al., 2013). In hot flash daily diaries, participants are asked to document their daily experiences of hot flashes as they occur by categorizing their symptom severity (mild, moderate, severe, and very severe). A participant's hot flash score is computed by adding the product of frequency x severity of hot flashes in each category.

SECONDARY OUTCOMES:
Hot Flash Related Daily Interference Scale | From enrollment to the end of treatment (week 6)
  Daily-life interference caused by hot flashes will be assessed using the Hot Flash Related Daily Interference Scale (HFRDIS; Carpenter et al., 2001). The HFRDIS is a 10-item scale that asks respondents to rate, on a 0-10 scale, the degree to which hot flashes interfere with various daily activities and overall enjoyment or quality of life. This measure has been shown to be valid and internally consistent, with an alpha of .96 (Carpenter et al., 2001). The HFRDIS will be administered at all measurement points (baseline and post-treatment).
Pittsburgh Sleep Quality Index | From enrollment to the end of treatment (week 6)
  The Pittsburgh Sleep Quality Index (PSQI; Buysse et al., 1989), a 19-item self-report questionnaire, will be administered to the participants across all three measurement points to evaluate sleep quality. Previous research demonstrates significant correlations between PSQI total scores and measures such as sleep onset latency, time spent awake after initial sleep onset, and total sleep time recorded by sleep diary and wrist actigraphy (Mollayeva et al., 2016). The PSQI will be administered at all measurement points (baseline and post-treatment).
Leeds Sleep Evaluation Questionnaire | End of treatment (week 6)
  The Leeds Sleep Evaluation Questionnaire (LSEQ; Parrott & Hindmarch, 1980) is a 10-item questionnaire that measures different dimensions of sleep and early morning behavior for the assessment of changes in sleep due to a treatment intervention. The scale was first introduced and validated in a clinical trial for the efficacy of temazepam for sleep quality and improved early morning behavior (Hindmach, 1975).
Hospital Anxiety Sub Scale | From enrollment to the end of treatment (week 6)
  Anxiety will be measured using the Hospital Anxiety Sub Scale (HADS; Zigmond & Snaith, 1983). The HADS-A is a 7-item self-report measure of patients' generalized anxiety over the past week. The HADS-A has shown internal consistency in previous studies with Cronbach's alphas ranging from .68-.93 and a mean of .83. It has also been shown to be correlated with other self-report measures of anxiety. The HADS-A will be administered at all measurement points (baseline and post-treatment).
Heart Palpitations | From enrollment to the end of treatment (week 6)
  Heart palpitations will be measured using a single-item baseline questionnaire. Women will be asked to rate their distress associated with "heart racing or pounding" in the past two weeks. The questionnaire will have five options, in which participants can select from "not at all" (0) to "extremely" (5). However, any indication of heart palpitations (ratings of 1 through 5) will be entered as a "yes" for palpitation distress in data analysis.
Perceived Stress Scale | From enrollment to the end of treatment (week 6)
  The Perceived Stress Scale (PSS; Cohen, 1983) is a 10-item scale that will be measuring the participants' stress before and after the intervention period. The scale provides the degree to which individuals find different situations of their lives to be unpredictable, uncontrollable, and overloaded, as well as measures the current levels of experienced stress. Items are scored on a scale from 0-4 with higher scores reflecting more perceived stress. This measure has been shown to be valid and internally consistent, with an alpha of .83 (Cohen, 1983). This scale will be administered at baseline and post-treatment.
App satisfaction and program ratings | End of treatment (week 6)
  Participants will be asked to rate their overall level of satisfaction with the app they used. A 10- point VAS scale (Wewers & Lowe, 1990) anchored with 0 "Completely Dissatisfied" to 10 "Completely Satisfied" will be given after 5 weeks of use. In order to assess participants' perceptions of the value of the app they receive, they will be asked, "How do you rate this app program overall regarding ease of use?" and "How do you rate this app program overall in regard to improving your hot flashes?" Responses will be given on a 10-point scale ranging from 1 (poor) to 10 (excellent) after completing 5 weeks of use.
Adherence | From enrollment to the end of treatment (week 6)
  Participants will be instructed to interact daily with the apps. Mindset Health will provide a log of user activity for data on adherence to the Evia app. In addition, the RAs will be inquiring on all participants' frequency of daily use during the weeks 1 through 5 phone calls. The research coordinator will closely monitor accrual and retention in addition to adverse events.
  Participants who drop out of the study will be contacted and given an opportunity to respond to an Exit Checklist to identify their reasons for dropping out.
Elkins Hypnotizability Scale-Clinical Form | End of treatment (week 6)
  Hypnotizability will be measured using the Elkins Hypnotizability Scale-Clinical Form (EHS-CF; Elkins, 2013). The EHS-CF is a standardized hypnotizability scale that is remotely administered using a Zoom call. The EHS-CF will be administered by a trained graduate student. The EHS-CF is highly correlated with longer measures of hypnotizability and has excellent validity and reliability in both a general and clinical population (Kekecs et al., 2016; Zimmerman et al., 2024). The EHS-CF takes approximately 20 minutes to administer and will be administered after the intervention. Those in the control condition will not complete the EHS-CF as they will not have any exposure to hypnosis (the EHS-CF involves a hypnotic induction).

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor University, Waco, Texas, United States

IPD SHARING:
Plan to Share IPD: No